CLINICAL TRIAL: NCT01993680
Title: A Monocentric Randomized, Controlled, Double Blind, Crossover Phase II Trial to Show Non-inferiority of the Effect of Pyridostigmine Bromide vs. Fludrocortisone on Symptoms of Autonomic Dysregulation in Parkinson's Disease
Brief Title: Orthostatic Dysregulation and Associated Gastrointestinal Dysfunction in Parkinson's Disease -Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Baumann (Other)
Responsible Party: Sponsor-Investigator, Christian Baumann, Professor dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KEK-ZH-NR. 2011-0358
Record Dates: First submitted 2012-04-27; First posted 2013-11-25 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Autonomic Disturbances in Parkinson's Disease
MeSH Terms: interventions — Pyridostigmine Bromide; Fludrocortisone; fludrocortisone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyridostigmine bromide (Experimental): 14 days of active treatment followed by 21 days wash out
  Interventions: Drug: Pyridostigmine bromide
- fludrocortisone (Active Comparator): 14 days of fludrocortisone treatment; 21 days wash out
  Interventions: Drug: fludrocortisone

INTERVENTIONS:
Drug: Pyridostigmine bromide — Drug doses during the trial:
  Pyridostigmine bromide: 30mg p.o. 1-1-1 to 2-2-2 given for 14 days
  Other Names: Mestinon
  Arms: Pyridostigmine bromide
Drug: fludrocortisone — drug dose during the trial Fludrocortisone: 0,1mg p.o. 1-0-0 to 2-0-0 given for 14 days
  Other Names: florinef
  Arms: fludrocortisone

SUMMARY:
Disabling symptoms of blood pressure dysregulation, impaired swallowing and digestion are common amongst Parkinson's patients. So far the exact pathophysiology for this is not fully understood. There are results from pathological analyses that the autonomic nervous system is also affected by the accumulation of alpha-Synuclein and that this might even happen in very early stages of the disease process (Qualman et al., 1984; Wakabayashi et al., 1989; Wakabayashi et al., 1990; Bloch et al., 2006).

Blood pressure dysregulation is a common autonomic symptom in Parkinson's patients and treatment - currently most often achieved with Fludrocortisone - often leads to supine hypertension (Plaschke et al., 1998; Braune et al., 1999; Magerkurth et al., 2005).

There are studies in patients with autonomic failure that indicate that Pyridostigmine bromide might be an alternative treatment option without causing disabling supine hypertension (Singer et al., 2003; Sandroni et al., 2005; Singer et al., 2006; Yamamoto et al., 2006).

Delayed gastric emptying is also an autonomic symptom associated with Parkinson's disease. By the elevation of the cholinergic tone with Pyridostigmine bromide the investigators also expect to alleviate symptoms of delayed gastric emptying and obstipation, possibly even facilitating the uptake of dopaminergic medication through the gut (Sadjadpour, 1983; Bharucha et al., 2008).

Therefore the investigators designed a monocentric randomized, controlled, double blind, crossover phase II trial to show non-inferiority of the effect of pyridostigmine bromide vs. fludrocortisone on symptoms of autonomic dysregulation in Parkinson's disease.

DETAILED DESCRIPTION:
In summary, investigators in recent years became more and more aware of the non-motor symptoms of PD and their impact on affected individuals. Therefore therapeutic strategies to ameliorate these symptoms are ever more needed. Sufficient clinical data for the treatment of symptoms of blood pressure dysregulation is still lacking. This study is aiming at closing this knowledge gap by comparing the efficacy and tolerability of a promising new agent, pyridostigmine bromide with the standard treatment, fludrocortisone.

The proposed target of pyridostigmine in this respect is at the autonomic ganglion in the efferent limb of the baroreflex. Via a reduction of acetylcholine breakdown the sympathetic ganglionic transmission increases upon orthostatic stress (Singer et al., 2006).

Via the same mechanism we aim to facilitate gastrooesophageal motility and gastric emptying: Both relaxation and contractibility of the oesophagus are known to be affected in PD patients as shown in a manometric study (Sung et al., 2010). Both relaxation and contractability are mainly influenced by nicotinergic and muscarinergic, cholinergic vagal efferents to the oesophagus (Chang et al., 2003). Via a reduction of acetylcholine breakdown we aim to increase the cholinergic tone and thereby normalize the reduced relaxation and contractibility.

We also intent to show that this faster gastric transit results in a faster absorption of Madopar into the bloodstream - we therefore will measure Levodopa and its metabolites during the first 60mins after ingestion of 125mg fast-release Madopar in serial venous blood samples via high-pressure liquid chromatography.

ELIGIBILITY:
Inclusion criteria:

* informed, written & formal consent for participation
* male / female subjects, aged 50-80 years
* PD patients (18 subjects with symptomatic orthostatic hypotension)

Exclusion criteria: - Antihypertensive treatment

* medication influencing gastrointestinal motility for at least the elimination half life of the drug
* medication interfering with blood-pressure regulation for at least the elimination half life of the drug
* significant systemic illness
* BMI <18 or >30kg/m2
* symptoms or a history of GI disease or surgery
* with any evidence of infectious disease
* evidence or history of drug or alcohol abuse
* diabetes mellitus

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2015-04 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in diastolic blood pressure drop on Schellong manoeuvre | 10min standing, 10 min supine
Changes in half emptying time t50 on 13C-sodium octanoate breath test | within 4h after test meal

SECONDARY OUTCOMES:
Efficacy of Pyridostigmine bromide | assess symptom severity for last 14 days
  central blood pressure, heart rate variability and pulse wave velocity
Efficacy of Pyridostigmine bromide | assess symptom severity for last 14 days
  Motor functions (UPDRS III), frequency and subjective quality of defecation, frequency and urgency of micturition, tremor severity (Whiget tremor scale);
Safety & Tolerability of Pyridostigmine bromide | assess symptom severity for last 14 days
  subjective assessment of sialorrhea, Hospital Anxiety and Depression Scale, Montreal Cognitive Assessment;

CONTACTS AND LOCATIONS:
Overall Officials: Christian Baumann, MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Singer W, Opfer-Gehrking TL, Nickander KK, Hines SM, Low PA. Acetylcholinesterase inhibition in patients with orthostatic intolerance. J Clin Neurophysiol. 2006 Oct;23(5):476-81. doi: 10.1097/01.wnp.0000229946.01494.4c. PMID 17016160
- [Background] Sandroni P, Opfer-Gehrking TL, Singer W, Low PA. Pyridostigmine for treatment of neurogenic orthostatic hypotension [correction of hypertension]--a follow-up survey study. Clin Auton Res. 2005 Feb;15(1):51-3. doi: 10.1007/s10286-005-0225-3. PMID 15768203
- [Derived] Schreglmann SR, Buchele F, Sommerauer M, Epprecht L, Kagi G, Hagele-Link S, Gotze O, Zimmerli L, Waldvogel D, Baumann CR. Pyridostigmine bromide versus fludrocortisone in the treatment of orthostatic hypotension in Parkinson's disease - a randomized controlled trial. Eur J Neurol. 2017 Apr;24(4):545-551. doi: 10.1111/ene.13260. Epub 2017 Feb 22. PMID 28224720